CLINICAL TRIAL: NCT01047241
Title: Nasal Administration of Sufentanil+Ketamine for Procedure-related Pain in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Danish University of Pharmaceutical Sciences (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Bettina Nygaard Nielsen, M.Sc. Pharm. sponsor contact person, Danish University of Pharmaceutical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201010; 2009-013801-33 (EudraCT Number)
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Pain
Keywords: Painful medical procedures
MeSH Terms: conditions — Pain | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intranasal sufentanil/ketamine (Experimental): Intranasal combination of sufentanil and ketamine. Dose of sufentanil 0.5 mcg/kg and ketamine 0.5 mg/kg, single dose.
  Interventions: Drug: Intranasal sufentanil/ketamine

INTERVENTIONS:
Drug: Intranasal sufentanil/ketamine — Nasal spray sufentanil+ketamine, 0,5 microg/kg sufentanil+0,5 mg/kg ketamine, single dose

SUMMARY:
The aim of the study is to investigate the absorption and clinical effect of nasal administration of an analgesic nasal spray containing sufentanil+ketamine for pain related to medical procedures in hospitalized children.

DETAILED DESCRIPTION:
The management of procedural pain in children ranges from physical restraint to pharmacological interventions. Pediatric formulations that permit accurate dosing, are accepted by children and a have a rapid onset of analgesia are lacking. The objectives were to investigate a pediatric formulation of intranasal sufentanil 0.5 mcg/kg and ketamine 0.5 mg/kg for procedural pain and to characterize the pharmacokinetic (PK) profile. Fifty children (≥10 kg) scheduled for a painful procedure were included in this prospective nonrandomized open-label clinical trial. Thirteen of these children had central venous access for drug assay sampling; enabling a compartmental PK analysis using nonlinear mixed-effects models. Pain intensity before and during the procedure was measured using age-appropriate pain scales. Heart rate, oxygen saturation and sedation were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents treated at the University Hospital, Rigshospital
* Painful medical procedure related to the patients treatment
* Patient and/or the parents must be able to understand and speak danish
* Negative pregnancy test for girls, when relevant
* Signed informed consent
* Only a light meals or no meals have been ingested 2 hours prior to inclusion

Exclusion Criteria:

* Allergy to sufentanil or ketamine
* Abnormal nasal cavity
* Have been treated with sufentanil and/or ketamine during the last 48 hours
* Nasal obstruction (rhinitis)

Ages: 1 Year to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2010-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steen W Henneberg, MD DMSc, Principal Investigator — Rigshospitalet, Denmark; Kjeld Schmiegelow, MD DMSc, Principal Investigator — Copenhagen University Hospital Righospitalet
Locations (1):
- Copenhagen University Hospital Rigshospitalet, Copenhagen, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Intranasal Sufentanil+Ketamine: Sufentanil, ketamine: Nasal spray sufentanil+ketamine, single dose
Period: Overall Study
Arm/Group | Intranasal Sufentanil+Ketamine
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intranasal Sufentanil+Ketamine
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.8 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 36
Weight [Mean (Standard Deviation); unit: kg] | 34.9 (20.1)
Height [Mean (Standard Deviation); unit: cm] | 138.4 (32.0)
Preprocedural pain intensity [Median (Inter-Quartile Range); unit: units on a scale] | 0.0 [0.0 to 2.0]

OUTCOME MEASURES:

1. Primary Outcome: Procedural Pain Intensity Score
Description: Children <5 years old were administered the FLACC (Face Leg Activity Cry Consolability) Scale (Range: 0-10, where 0 is no pain and 10 is worst pain). Children >= 5 years but < 8 years old were administered the Visual analog scale modified with six faces by Wong-Baker (Wong-Baker Faces Pain Rating Scale) (Range: 0-10, where 0 is no pain and 10 is worst pain). Children >= 8 years old were administered a Visual Analog Scale (Range: 0-10, where 0 is no pain and 10 is worst pain).
Time Frame: Pain assessment during painful medical procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Intranasal Sufentanil/Ketamine: Sufentanil/ketamine: Nasal spray containing a combination of sufentanil and ketamine. Dose sufentanil 0.5 micg/kg and ketamine 0.5 mg/kg, single dose
Arm/Group | Intranasal Sufentanil/Ketamine
Number analyzed (Participants) | 50
units on a scale | 3.1 [2.0 to 4.9]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Sufentanil and Ketamine
Time Frame: Time= 5-60 min after administration of the investigational medical product
Measure: Mean (Standard Deviation); unit: mcg/L
Groups:
- Intranasal Sufentanil/Ketamine: Sufentanil/ketamine: Nasal spray containing a combination of sufentanil and ketamine. Dose sufentanil 0.5 micg/kg and ketamine 0.5 mg/kg, single dose Pharmacokinetic analysis: 13 children enrolled
Arm/Group | Intranasal Sufentanil/Ketamine
Number analyzed (Participants) | 12
mcg/L
  Cmax sufentanil | 0.042 (0.005) [0.151 to 0.277]
  Cmax ketamine | 102 (11)

3. Secondary Outcome: Sedation Score (UMSS)
Description: University of Michigan Sedation Score (UMSS) (0-4, 0 "awake and alert", 4 "unarousable")
Time Frame: Time= 0-70 min. after drug administration
Measure: Median (Full Range); unit: units on a scale
Groups:
- Intranasal Sufentanil/Ketamine: Sufentanil/ketamine: Nasal spray containing sufentanil/ketamine. Dose sufentanil 0.5 mcg/kg and ketamine 0.5 mg/kg, single dose.
Arm/Group | Intranasal Sufentanil/Ketamine
Number analyzed (Participants) | 50
units on a scale | 0 [0 to 2]

4. Secondary Outcome: Acceptance of Intranasal Administration
Description: Asking the children (parents for preverbal children) if they would like to receive this treatment again in a similar situation rather than analgesic suppositories, tablets, oral solutions, or injections?
Time Frame: Immediately after the procedure
Measure: Number; unit: percentage of participants
Groups:
- Intranasal Sufentanil/Ketamine: Sufentanil/ketamine: Nasal spray containing a combination of sufentanil and ketamine. Dose sufentanil 0.5 mcg/kg and ketamine 0.5 mg/kg, single dose.
Arm/Group | Intranasal Sufentanil/Ketamine
Number analyzed (Participants) | 50
percentage of participants | 47

5. Primary Outcome: Bioavailability of Sufentanil and Ketamine
Time Frame: Time= 5-60 min after administration of the investigational medical product
Measure: Mean (Standard Error); unit: percentage bioavailable
Arm/Group | Intranasal Sufentanil/Ketamine
Number analyzed (Participants) | 12
percentage bioavailable
  Bioavailability sufentanil | 24.6 (18.5)
  Bioavailability ketamine | 35.8 (15.4)

6. Primary Outcome: Time to Maximum Plasma Concentrations (Tmax) Sufentanil and Ketamine
Time Frame: Time=5-60 min after administration of investigational medicinal product
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intranasal Sufentanil/Ketamine
Number analyzed (Participants) | 12
minutes
  Tmax sufentanil | 13.8 (1.7)
  Tmax ketamine | 8.5 (1.5)

ADVERSE EVENTS:
Arm/Group | Intranasal Sufentanil+Ketamine
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 2/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intranasal Sufentanil+Ketamine (N=50)
Vomiting (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes